CLINICAL TRIAL: NCT04502394
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of KRT-232 in Combination With Acalabrutinib in Subjects With Relapsed/Refractory Diffuse Large B-cell Lymphoma or Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Safety and Efficacy of KRT-232 in Combination With Acalabrutinib in Subjects With R/R DLBCL or R/R CLL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-111
Record Dates: First submitted 2020-07-27; First posted 2020-08-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B Cell Lymphoma; Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
Keywords: navtemadlin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; acalabrutinib

STUDY DESIGN:
Intervention Model Description: An Open-label, Phase 1b/2 Study of KRT-232 in combination with acalabrutinib in Subjects with B-cell Non-Hodgkin Lymphoma
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (R/R DLBCL) (Experimental): KRT-232 will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle.
  Acalabrutinib at 100 mg twice a day (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: acalabrutinib
- Cohort 2 (R/R CLL) (Experimental): KRT-232 will be administered orally, once daily (QD), on days 1-7 in a 28-day cycle.
  Acalabrutinib at 100 mg twice a day (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: acalabrutinib

INTERVENTIONS:
Drug: KRT-232 — KRT-232 is an experimental MDM2 inhibitor anticancer drug taken by mouth
Drug: acalabrutinib — acalabrutinib is a BTK inhibitor anticancer drug taken by mouth
  Other Names: ACP-196

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, combined with acalabrutinib for the treatment of adults with Diffuse Large B-Cell Lymphoma and Chronic Lymphocytic Leukemia. Participants must be relapsed/refractory (having failed prior therapy)

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Confirmed diagnosis of TP53wt DLBCL (WHO); R/R DLBCL after at least 2 prior lines of treatment or 1 prior for patients who are ineligible for stem cell transplant
* Cohort 2: Confirmed diagnosis of TP53wt CLL (iwCLL); R/R CLL after at least 1 prior line of treatment
* ECOG 0 to 2
* Adequate hematologic, hepatic, and renal functions.

Exclusion Criteria:

* Prior treatment with any MDM2 inhibitor
* Prior treatment with any BTK inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Primary Objective Phase 1b:To determine the KRT-232 maximum tolerated dose/ maximum administered dose (MTD/MAD) and recommended Phase 2 Dose (RP2D) in combination with acalabrutinib in subjects with R/R DLBCL or R/R CLL | 56 Days
  Endpoint/Outcome Measures: Dose-limiting toxicities will be used to establish the MTD/MAD of KRT-232 in combination with acalabrutinib. The Safety Review Committee will determine the RP2D based on safety data of the combination of KRT-232 and acalabrutinib.
Primary Objective Phase 2: Cohort 1: To determine the complete response (CR) | 1 Year
  Endpoint/Outcome Measures: Cohort 1: The proportion of subjects with CR as assessed by investigators per the Lugano Classification.
Primary Objective Phase 2: Cohort 2: To determine the rate of CR/complete remission with incomplete hematologic recovery (CRi) rate in R/R CLL | 1 Year
  Endpoint/Outcome Measures: Cohort 2: The proportion of subjects with CR/CRi as assessed by investigators per iwCLL Response Criteria.

SECONDARY OUTCOMES:
Phase 1b Secondary Objective: Pharmacokinetic (PK) profile | Baseline, 1, 2, 4, 6 and 24 hours post dose on days 1 and 2 of cycle 1 (each cycle is 28 days); Baseline and 2 hours post dose on day 1 and 24 hours post dose on day 8 of cycle 2
  Endpoint/Outcome Measures: Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameter from a single dose will be estimated maximum concentration (Cmax).
Phase 1b Secondary Objective: Pharmacokinetic (PK) profile | Baseline, 1, 2, 4, 6 and 24 hours post dose on days 1 and 2 of cycle 1 (each cycle is 28 days); Baseline and 2 hours post dose on day 1 and 24 hours post dose on day 8 of cycle 2
  Endpoint/Outcome Measures: Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameters from a single dose will be area under the curve (AUC).
Phase 1b Secondary Objective: Pharmacokinetic (PK) profile | Baseline, 1, 2, 4, 6 and 24 hours post dose on days 1 and 2 of cycle 1 (each cycle is 28 days); Baseline and 2 hours post dose on day 1 and 24 hours post dose on day 8 of cycle 2
  Endpoint/Outcome Measures: Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameters from a single dose will be half-life (T1/2).
Phase 1b Secondary Objective: Pharmacokinetic (PK) profile | Baseline, 1, 2, 4, 6 and 24 hours post dose on days 1 and 2 of cycle 1 (each cycle is 28 days); Baseline and 2 hours post dose on day 1 and 24 hours post dose on day 8 of cycle 2
  Endpoint/Outcome Measures: Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameter from a single dose will be apparent clearance.
Phase 1b Secondary Objective: Pharmacokinetic (PK) profile | Baseline, 1, 2, 4, 6 and 24 hours post dose on days 1 and 2 of cycle 1 (each cycle is 28 days); Baseline and 2 hours post dose on day 1 and 24 hours post dose on day 8 of cycle 2
  Endpoint/Outcome Measures: Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameters from a single dose will be apparent volume of distribution using non-compartmental or compartmental PK methods with the software WinNonlin.
Phase 2 Secondary Objective: Cohort 1 (R/R DLBCL): To determine the overall response rate (ORR) for R/R DLBCL subjects. | 2 Years
  Endpoint/Outcome Measures: The proportion of subjects who achieve a partial response (PR) or better at any time point while on study.
Phase 2 Secondary Objective: Cohort 2 (R/R CLL): To determine the ORR for R/R CLL subjects | 2 Years
  Endpoint/Outcome Measures: The proportion of subjects who achieve a PR or better at any time point while on study, as assessed by iwCLL Response Criteria

CONTACTS AND LOCATIONS:
Locations (45):
- United States (4):
  - Goshen Center for Cancer Care, Goshen, Indiana
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Eastern Health - Box Hill Hospital, Box Hill
  - Barwon Health, Geelong
  - Royal Perth Hospital, Perth
- Belgium (3):
  - Antwerp University Hospital (UZA), Edegem
  - Jessa Ziekenhuis, Hasselt
  - University Hospital (UZ) Leuven, Leuven
- Czechia (3):
  - Fakultni Nemocnice Hradec Kralove, Nový Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (3):
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Centre Henri Becquerel, Rouen
  - CHRU de Tours - Hôpital Bretonneau, Tours
- Italy (6):
  - Centro Riferimento Oncologico - Aviano, Aviano
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Poland (6):
  - Copernicus PL Sp. z o.o., Wojewodzkie Centrum Onkologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Oddzial w Gliwicach - Klinika Transplantacji Szpiku i Onkohematologii, Gliwice
  - Pratia MCM Krakow, Krakow
  - Szpital Uniwersytecki Krakow - Oddzial Kliniczny Hematologii, Krakow
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (5):
  - Hospital de Braga, Braga
  - Centro Hospitalar Universitario de Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Champalimaud Cancer Center, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho EPE, Vila Nova de Gaia
- South Korea (6):
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- United Kingdom (4):
  - St James's University Hospital, Leeds
  - King's College Hospital, London
  - Royal Marsden Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton